CLINICAL TRIAL: NCT03907956
Title: Efficacy of Dry Needling With the Fascial Winding Technique in the Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Jordi Gascon-Garcia, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JGascon-Garcia
Record Dates: First submitted 2019-03-18; First posted 2019-04-09 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: physiotherapy; carpal tunnel syndrome; myofascial pain syndrome; dry needling
MeSH Terms: conditions — Carpal Tunnel Syndrome; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: The study is a randomized single-blind clinical trial (RCT).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Assignment to groups. To the extent that the sample is recruited, subjects will be randomly distributed into two groups (intervention and control) using a software-generated randomization system. Each subject will be assigned a numbered, sealed and opaque envelope where their inclusion in the intervention or control group will be specified.
  The evaluating staff will be blinded to the assignment to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): The subjects included in the intervention group will be treated with Dry Needling with Fascial Winding Technique according to the original Four-Pole Carpal Dry Needling approach, which has already been validated recently by means of a first ultrasound study.
  Interventions: Other: Dry Needling with Fascial Winding Technique
- CONTROL (No Intervention): The individuals of the control group will remain within the normal course of their waiting list status for CTS surgery, without receiving any extraordinary treatment to what is normally practiced in this situation.

INTERVENTIONS:
Other: Dry Needling with Fascial Winding Technique — For placement of Dry Needling (DN) needles with Fascial Winding Technique (FWT) according to the Four-pole Carpal Dry Needling (FCDN) approach model, only anatomical references are used, in all cases from a carpal ventral approach. The needles used are the Chinese type with silver handle and guide tube, measuring 25x0.30 mm., Agupunt® brand. Four needles are placed, at the level of the bones: scaphoid, pisiform, trapezius and hamate. The four needles follow an oblique direction, always on the back and looking for the midline of the center of the carpal tunnel, with an inclination of approximately 45º, both in the cranio-caudal and medial-lateral directions. In each of the needles, it deepens until it reaches a firm elastic stop, attributable to the Transverse Carpal Ligament. Next, the FWT is applied to each of the needles, consisting of rotating them in the same direction until you feel the final stop of the "needle grasp".
  Arms: INTERVENTION

SUMMARY:
So far there are studies that report the benefits of physiotherapy treatment in carpal tunnel syndrome, but none on the treatment of dry needling. Recently, an ultrasound validation study has been published in which the results indicate that the application of dry needling with "fascial winding technique" in the carpal tunnel, following the "four-pole carpal dry needling" model, is valid for reaching and traction of the transverse carpal ligament. Stretching over this ligament could lead to new therapeutic possibilities for dry needling at this level. The objective of this project is to demonstrate the clinical efficacy of this technique in patients affected by carpal tunnel syndrome, determining the proportion of patients who can be avoided surgery, and quantifying the improvement in the clinic related to pain, strength and functionality of the hand and the median nerve.

The study is a randomized clinical trial on a sample of 86 patients diagnosed with carpal tunnel syndrome, who have been prescribed surgery at this level. The degree of involvement of the median nerve will be mild or moderate, according to electromyographic results. The dry needling with fascial winding technique will be applied to the intervention group following the model of "four-pole carpal dry needling" during a period of 6 weeks, at the rate of one weekly session. The control group will remain within the normal course of their waiting list status for STC surgery, without receiving any extraordinary treatment to what is normally practiced in this situation. The main variables contemplated are: need for surgery at the end of the study, level of involvement of the median nerve (according to electromyographic result), transverse area of the median nerve at the entrance of the carpal tunnel and relationship between the area of the median nerve at the wrist and the forearm (both recorded by ultrasound study), pain intensity (using visual analog scale), symptom intensity, functional capacity and quality of life (according to the Boston Carpal Tunnel Questionnaire), and degree of muscular strength to the grip manual and digital.

DETAILED DESCRIPTION:
INTRODUCTION:

Dry Needling (DN) is an invasive technique widely used in the Physiotherapy field, on which numerous studies have recently been published. The vast majority of these studies focus on the action of DN on the muscular element: the well-known myofascial trigger points. According to what Dunning proposed in 2014, it should not ignore and/or underestimate its action on the connective-fascial tissue, the other aspect of a single, unique and indivisible functional whole: the myofascia.

In the field of acupuncture, numerous studies have been conducted to determine the role played by the fascia in the therapeutic phenomenon that begins when working with a needle. Among these, mention in particular the studies of Dr. H. M. Langevin, pioneers in the contribution of scientific evidence to the phenomenon known as "needlegrasp". When the acupuncture needle (the same as the one used in DN) is rotated, the fascial connective tissue winds around to the point where it is fastened and trapped.

With the intention of demonstrating the benefit of treatment with DN on connective-fascial tissue, the investigators present this research project. In the same, it is proposed to apply DN in a pathology such as carpal tunnel syndrome (CTS), in which surgical treatment is currently considered principally.

There are previous studies that describe the benefits of physiotherapy treatment in the CTS, but none on the treatment of DN. Recently, it has been validated using ultrasound image how DN needles, applied following the original model proposed and described as "four-pole carpal dry needling" (FCDN), reach the transverse carpal ligament (TCL) in 93.1%. In turn, if these needles are manipulated in the form of unidirectional rotation, named in this work as "fascial winding technique" (FWT), a traction-stretching of this ligament can be observed via ultrasound. It was possible to observe in 80.6% of the occasions. The results obtained indicate that DN with FWT in the carpal tunnel (CT), following the FCDN model, is valid to reach and traction the TCL. Similarly, the same study also shows this treatment as safe in terms of not injuring the median nerve and/or the ulnar artery. The level of pain and/or superficial bleeding produced is very slight and only at the time of performing the technique, without causing painful discomfort or residual bruising.

In affected patients with CTS there is a decrease in the sliding movement of the median nerve with respect to the TCL, located just above it. If, as has already been verified, a traction-stretching of the TCL can be performed using the DN technique with FWT applied according to the FCDN model, a relaxation of the tension and flexibility in this same ligament can also be achieved . It is logical to think that this decrease in the tension of the TCL leads to an improvement in the sliding movement of the median nerve, restricted in patients with CTS. On the other hand, this relaxation of the TCL (one of the walls of the case that forms the CT) could also lead to a decrease in the pressure existing inside the tunnel, thus decreasing the compression on the median nerve, established as one of the main causes of the symptoms of sensory and motor disturbance in these patients.

If it is possible to demonstrate the clinical efficacy of DN treatment with FWT in patients with CTS, important benefits will be achieved. In the first place, a new therapeutic tool would be provided, full of competence for the physiotherapist, in the treatment of this pathology. In addition, the combination of this treatment with other medical and physiotherapeutic types already existing could increase the therapeutic benefits for patients with CTS. It is even contemplated that it is shown to be effective enough to be considered as an alternative to surgery in cases of mild or moderate medium nerve involvement, thus avoiding all the risks and possible complications that this entails. For all this, the economic burden derived from the current treatment in these patients, as well as the time of convalescence and/or sick leave, would be significantly reduced.

HYPOTHESIS:

Dry needling with fascial winding technique applied in patients with carpal tunnel syndrome in a level of mild or moderate median nerve involvement, avoids surgery, at this level, to a significant proportion of patients with indication of it.

OBJECTIVES:

PRINCIPAL:

o To determine the proportion of patients with carpal tunnel syndrome and level of mild or moderate median nerve involvement in which the application of dry needling with a fascial winding technique avoids surgery at this level.

ESPECIFIC:

* To determine the improvement in the clinic related to pain, strength and functionality of the hand and the median nerve, in patients with carpal tunnel syndrome treated with dry needling with fascial winding technique.
* Determine if there are adverse or undesirable effects when applying dry needling with fascial winding technique in patients with carpal tunnel syndrome and, if so, specify what they are and how often they occur. In this same line, the intensity of pain associated with the application of the "four-pole carpal dry neeling" approach will be determined.

METHODOLOGY:

The study is a randomized single-blind clinical trial (RCT).

Sample. The individuals of the sample will be recruited by sampling of consecutive cases of the Orthopedic Surgery and Traumatology Service of Hospital de Bellvitge, once the carpal tunnel surgery is considered indicated.

Sample size:

The calculation of the number of individuals required has been made taking into account that currently the percentage of success of open surgery ranges between 70-98%, so it is expected to avoid such surgery at a percentage of 84 ± 12.5%. Setting a power of 80% and a level of significance of 5% in the ratio comparison formula for cases of bioequivalence, we obtain that the sample size is 34 individuals per group. Assuming a maximum loss percentage of 20% it will be necessary to recruit 43 individuals per group.

Assignment to groups. To the extent that the sample is recruited, subjects will be randomly distributed into two groups (intervention and control) using a software-generated randomization system. Each subject will be assigned a numbered, sealed and opaque envelope where their inclusion in the intervention or control group will be specified. The evaluating staff will be blinded to the assignment to the groups.

STATISTICAL ANALYSIS OF THE DATA:

First, a descriptive analysis of the sociodemographic characteristics (age, sex and profession) and anthropometric characteristics (BMI, wrist perimeter, dominant hand) for each of the groups and for all response variables (EMG, CSA-M , WF-R, pain intensity, BCTQ, muscle strength of grip, and intensity of pain that causes the FCDN approach model) for each of the groups and for each of the assessments. For this, the percentage for the qualitative variables and the mean and standard deviation for the quantitative ones will be calculated.

Secondly, the evolution of each one of the response variables will be evaluated and they will be compared between both groups with a two-factor ANOVA test and with repeated measures. The level of significance set is 5%. The statistical analysis will be carried out with the SPSS 21.0 software.

ETHICAL ASPECTS:

Note that this project complies with the principles established in the Declaration of Helsinki, and will be submitted for approval to the Clinical Research and Ethics Committee of Bellvitge Hospital.

All participating subjects will sign an informed consent, with free and voluntary acceptance of participation in the study.

ELIGIBILITY:
Inclusion Criteria:

The study population are individuals with a clinical and electromyographic diagnosis of CTS, and levels of mild median nerve involvement (focal demyelination without axonal degeneration) or moderate (focal demyelination with sensory but non-motor axonal degeneration) according to electromyogram (EMG).

Exclusion Criteria:

Will not be included those subjects with previous surgery in the CT, to whom the involvement of the median nerve is attributable to another type of neuropathy (diabetic, uraemic, deficiency, ...), to those who present a previous pain in the region, attributable to arthritis and not to CTS, to individuals suffering from fibromyalgia and/or chronic pain syndrome, to those who suffer from aversion or phobia to needles, to pregnant patients, to those with intellectual disability to understand the procedure, methodology and object of the study (mental, psychiatric disorders, low level of IQ, ...), and/or those patients who show little collaboration to the correct performance of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
The need to continue performing surgery for carpal tunnel syndrome. | Before the start of treatment (week 0) and after 6 weeks of the end of treatment (week 12), in all the subjects participating in the study
  According to the tests carried out and under medical criteria, at the end of the study will be assessed the need to continue performing surgery at this level for each of the individuals who participated in the study.

SECONDARY OUTCOMES:
Level of involvement of the median nerve, registered by EMG. | Before the start of treatment (week 0) and after 6 weeks of the end of treatment (week 12), in all the subjects participating in the study
  The EMG is a totally objective and validated test to assess the degree of involvement of the median nerve, being considered as the "gold standard" for the diagnosis of CTS
Cross sectional area of the median nerve at the wrist tunnel (CSA-M) | Before the start of treatment (week 0) and after 6 weeks of the end of treatment (week 12), in all the subjects participating in the study
  Registered by ultrasound study. It has recently been shown that there is a relationship between the transverse area of the median nerve in the wrist and the severity of the CTS (39, 40). It is considered that such measurements can be complementary to diagnose the CTS and determine its severity.
Wrist-forearm relationship (WF-R) | Before the start of treatment (week 0) and after 6 weeks of the end of treatment (week 12), in all the subjects participating in the study
  Registred by ultrasound study. The study of the relationship between the area of the median nerve in the wrist and the forearm (WF-R) is contemplated to minimize the possible effect of the variability in the population with respect to the absolute results of the CSA-M values, considering its sensitivity higher than that of WF-R according to some authors
Intensity of pain, collected and measured with a Visual Analogue Scale (VAS). | For Intervention group: Before the start of treatment (week 0), every two weeks (weeks 2, 4, 6 and 8) and after 6 weeks of the end of treatment (week 12). For Control group: week 0, week 6 and wek 12
  Previous studies have demonstrated the validity of VAS in pain measurement. The patient will mark his level of pain in a ruler numbered from 0 to 10 cm, where 0 is absence of pain and 10 unbearable pain. This assessment will include: pain that presents just at the time of performing the VAS, pain in the last 24 hours, and pain presented in the last week.
Boston Carpal Tunnel Questionare (BCTQ) | For Intervention group: Before the start of treatment (week 0), every two weeks (weeks 2, 4, 6 and 8) and after 6 weeks of the end of treatment (week 12). For Control group: week 0, week 6 and wek 12
  Intensity of symptoms, functional capacity and quality of life. Specifically designed and validated for the diagnosis of CTS (47, 48). The BCTQ contains questions regarding pain, paresthesia and hand functionality. It is reproducible, validated in Spanish and with internal consistency, capable of responding to clinical and transcultural changes.
Muscular strength to manual and digital grasping. | For Intervention group: Before the start of treatment (week 0), every two weeks (weeks 2, 4, 6 and 8) and after 6 weeks of the end of treatment (week 12). For Control group: week 0, week 6 and wek 12
  Collection and measurement with a dynamometry test. The data is measured using a Jamar hydraulic dynamometer, validated in previous studies (49-51), and which expresses the isometric strength of hand grip.
Visual Analogue Scale (VAS) for Intensity of pain caused by the Four Carpal Dry Needling (FCDN) approach model. | Only in the Intervention group: in the weeks 2, 4 and 6.
  The patient will mark his level of pain in a ruler numbered from 0 to 10 cm, where 0 is absence of pain and 10 unbearable pain. Data will be collected just after placing and manipulating the needles, as well as after removing them after 10 minutes.
Positive Clinical Diagnosis of CTS | Before the start of treatment (week 0) and after 6 weeks of the end of treatment (week 12), in all the subjects participating in the study
  According to the criteria established by the American Academy of Orthopedic Surgeons (AAOS), we understand a positive clinical diagnosis of CTS when the patient presents a sensitive clinic of pain in the hand and/or paresthesias in the sensory distribution of the median nerve, and/or motor clinic with loss of strength of the thenar muscles, which can be objectified with atrophy of them. In addition to this sensitive and motor clinical presentation, it is advisable to establish a clinical diagnosis of CTS when the positive result of one or several of these signs or provocation test is associated: Phalen test, Tinel's sign, compression test of the median nerve, and/or Flick sign.
Adverse or unwanted effects. | Only in the Intervention group: in the weeks 2, 4, 6 , 8 and 12.
  Data will be collected regarding the increase and duration of post-treatment pain, as well as the appearance of other possible complications or unwanted effects. A document will be provided to record the appearance of these possible adverse or undesirable effects derived from the applied treatment.

OTHER OUTCOMES:
Age | Before the start of treatment (week 0)
  The age of the individuals included in the sample will be collected.
Sex | Before the start of treatment (week 0)
  The sex of the individuals included in the sample will be collected.
Profession | Before the start of treatment (week 0)
  The profession of the individuals included in the sample will be collected.
Body Mass Index (BMI) | Before the start of treatment (week 0)
  The BMI of the individuals included in the sample will be collected.
Wrist circumference | Before the start of treatment (week 0)
  The Wrist circumference, in cm., of the individuals included in the sample will be collected.
Dominant hand | Before the start of treatment (week 0)
  The dominant hand of the individuals included in the sample will be collected.
Medication. | For Intervention group: Before the start of treatment (week 0), every two weeks (weeks 2, 4, 6 and 8) and after 6 weeks of the end of treatment (week 12). For Control group: week 0, week 6 and wek 12
  Data will be collected regarding whether the individuals included in the sample have taken medication and, if so, what type, both in the last week before starting treatment and during the performance of the same.
Existence of cervical pain. | Before the start of treatment (week 0) and after 6 weeks of the end of treatment (week 12), in all the subjects participating in the study
  It will be registered if the individuals included in the sample suffer cervical pain and, if so, from how long.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Gascon-Garcia, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
For the time being it is expected to analyze the data obtained for the elaboration of the study that we present. It is to be determined if in the future these data can be used for other studies.